CLINICAL TRIAL: NCT01623557
Title: A Phase I/IIa Sporozoite Challenge Study to Assess the Protective Efficacy of Two Prime-Boost Malaria Vaccine Candidates: ChAd63 and MVA Encoding ME-TRAP and the Same Viral Vectors Encoding CS
Brief Title: A Challenge Study to Assess the Protective Efficacy of Two Malaria Vaccine Candidates
Acronym: VAC045
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: VAC045
Record Dates: First submitted 2012-05-16; First posted 2012-06-20 (Estimated); Last update posted 2015-02-16 (Estimated); Status verified 2015-02

CONDITIONS: Plasmodium Falciparum Malaria
Keywords: Malaria; Vaccine; Plasmodium; falciparum
MeSH Terms: conditions — Malaria, Falciparum; Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1: ChAd63-MVA CS (Active Comparator): 1 dose of ChAd63 CS 5 x 10^10 vp intramuscularly and 1 dose MVA CS 2 x 10^8 pfu intramuscularly 8 weeks later.
  Interventions: Biological: ChAd63-MVA CS; Other: Controlled Human Malaria Infection Administered by Mosquito Bite
- Group 2: ChAd63-MVA ME-TRAP (Active Comparator): 1 dose of ChAd63 ME-TRAP 5 x 10^10 vp intramuscularly and 1 dose MVA ME-TRAP 2 x 10^8 pfu intramuscularly 8 weeks later.
  Interventions: Biological: ChAd63-MVA ME-TRAP; Other: Controlled Human Malaria Infection Administered by Mosquito Bite
- Group 3: Unvaccinated Infectivity Controls (Active Comparator)
  Interventions: Other: Controlled Human Malaria Infection Administered by Mosquito Bite

INTERVENTIONS:
Biological: ChAd63-MVA CS — 1 dose of ChAd63 CS 5 x 10^10 vp intramuscularly and 1 dose MVA CS 2 x 10^8 pfu intramuscularly 8 weeks later.
  Arms: Group 1: ChAd63-MVA CS
Biological: ChAd63-MVA ME-TRAP — 1 dose of ChAd63 ME-TRAP 5 x 10^10 vp intramuscularly and 1 dose MVA ME-TRAP 2 x 10^8 pfu intramuscularly 8 weeks later.
  Arms: Group 2: ChAd63-MVA ME-TRAP
Other: Controlled Human Malaria Infection Administered by Mosquito Bite — Approximately 3 weeks post MVA dosing

SUMMARY:
This study aims to assess the safety and effectiveness of four new candidate malaria vaccines; ChAd63 CS, ChAd63 ME-TRAP, MVA CS & MVA ME-TRAP. These vaccines consist of viruses (ChAd63 and MVA) which have been genetically modified so (i) they cannot replicate in humans and (ii) they include parts of the malaria parasite; Plasmodium falciparum (CS and ME-TRAP). The hope is that these vaccines will induce immune responses in vaccinees that are able to prevent malaria.

This proposed study will compare how effective ChAd63-MVA CS is at preventing malaria infection in UK volunteers following malaria challenge compared to ChAd63-MVA ME-TRAP.

The study will be conducted at the University of Oxford's Centre for Clinical Vaccinology and Tropical Medicine (CCVTM), Oxford, UK and the Wellcome Trust Clinical Research Facility in Southampton, UK. The malaria challenge will take place at the insectary at Imperial College (Infection and Immunity Section) in London, UK.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18 to 45 years.
* Able and willing (in the Investigator's opinion) to comply with all study requirements.
* Willing to allow the investigators to discuss the volunteer's medical history with their General Practitioner.
* Women only: Must practice continuous effective contraception for the duration of the study.
* Agreement to refrain from blood donation during the course of the study and for at least 3 years after the end of their involvement in the study.
* Written informed consent to participate in the trial.
* Reachable (24/7) by mobile phone during the period between CHMI and completion of antimalarial treatment.
* Willingness to take a curative anti-malaria regimen following CHMI.
* For volunteers not living in Oxford: agreement to stay in a hotel room close to the trial centre during a part of the study (from at least day 6.5 post mosquito bite until anti-malarial treatment is completed).
* Answer all questions on the informed consent quiz correctly.

Exclusion Criteria:

* History of clinical malaria (any species).
* Travel to a malaria endemic region during the study period or within the preceding six months with significant risk of malaria exposure.
* Use of systemic antibiotics with known antimalarial activity within 30 days of CHMI (e.g. trimethoprim-sulfamethoxazole, doxycycline, tetracycline, clindamycin, erythromycin, fluoroquinolones and azithromycin)
* Receipt of an investigational product in the 30 days preceding enrolment, or planned receipt during the study period.
* Prior receipt of an investigational malaria vaccine or any other investigational vaccine likely to impact on interpretation of the trial data.
* Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (inhaled and topical steroids are allowed).
* Use of immunoglobulins or blood products within 3 months prior to enrolment.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine (e.g. egg products, Kathon) or malaria infection.
* Any history of anaphylaxis post vaccination.
* History of clinically significant contact dermatitis.
* History of sickle cell anaemia, sickle cell trait, thalassemia or thalassemia trait or any haematological condition that could affect susceptibility to malaria infection.
* Pregnancy, lactation or intention to become pregnant during the study.
* Contraindications to the use of all three proposed anti-malarial medications; Malarone, Riamet and Chloroquine.
* History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ).
* History of serious psychiatric condition that may affect participation in the study.
* Any other serious chronic illness requiring hospital specialist supervision.
* Suspected or known current alcohol abuse as defined by an alcohol intake of greater than 42 units every week.
* Suspected or known injecting drug abuse in the 5 years preceding enrolment.
* Seropositive for hepatitis B surface antigen (HBsAg).
* Seropositive for hepatitis C virus (antibodies to HCV) with positive PCR for hepatitis C at screening.
* An estimated, ten year risk of fatal cardiovascular disease of ≥5%, as estimated by the Systematic Coronary Risk Evaluation (SCORE) system.76
* Positive family history in 1st and 2nd degree relatives < 50 years old for cardiac disease.
* Volunteers unable to be closely followed for social, geographic or psychological reasons.
* Any clinically significant abnormal finding on biochemistry or haematology blood tests, urinalysis or clinical examination.
* Any other significant disease, disorder or finding which may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2012-04; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
The effectiveness of ChAd63-MVA CS and ChAd63-MVA ME-TRAP at preventing malaria infection | Up to 30 days post challenge
  Comparison of the number of individuals who develop malaria infection between vaccinees and unvaccinated control volunteers.

SECONDARY OUTCOMES:
The safety and immunogenicity of ChAd63-MVA CS and ChAd63-MVA ME-TRAP | up to 7 months post first vaccination
  The safety of the vaccine regimens will be assessed by analysing actively and passively collected data from clinical review of volunteers and laboratory measurements.
  The ability of the vaccines to induce malaria-specific immune responses (immunogenicity) will be assessed by the following laboratory tests;
  (A) Interferon gamma ELISPOT. (B) Flow cytometry to measure T cell responses
  Other laboratory investigations including microarray analysis may be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Adrian V S Hill, MD, Principal Investigator — University of Oxford
Locations (3):
- United Kingdom (3):
  - Centre for Clinical Vaccinology and Tropical Medicine, Oxford, Oxfordshire
  - Infection and Immunity Section, Imperial College of Science, Technology and Medicine, London
  - Wellcome Trust CRF, Southampton General Hospital, Southampton

REFERENCES:
- [Derived] Hodgson SH, Ewer KJ, Bliss CM, Edwards NJ, Rampling T, Anagnostou NA, de Barra E, Havelock T, Bowyer G, Poulton ID, de Cassan S, Longley R, Illingworth JJ, Douglas AD, Mange PB, Collins KA, Roberts R, Gerry S, Berrie E, Moyle S, Colloca S, Cortese R, Sinden RE, Gilbert SC, Bejon P, Lawrie AM, Nicosia A, Faust SN, Hill AV. Evaluation of the efficacy of ChAd63-MVA vectored vaccines expressing circumsporozoite protein and ME-TRAP against controlled human malaria infection in malaria-naive individuals. J Infect Dis. 2015 Apr 1;211(7):1076-86. doi: 10.1093/infdis/jiu579. Epub 2014 Oct 21. PMID 25336730